CLINICAL TRIAL: NCT05947773
Title: Effect of Robotic Treatments on Motor Functions in Subacute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Head of Department, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB/2022/02
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: robotic; stroke; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robotically treated patient (Experimental): They performed training with a robot 15 times over 3 weeks.
  Interventions: Other: Learning to walk with a robot
- Walking training (Experimental): Walking exercises were performed without a robot.
  Interventions: Other: Walking group
- Control group (Experimental): Physiotherapy treatment was carried out by the patients.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Learning to walk with a robot — The patients completed a 1-hour learning to walk program using a soft exoskeleton. The protocol includes several difficult parts of the walk. (Walking protocol)
  Other Names: ROB
  Arms: Robotically treated patient
Other: Walking group — The walking protocol was performed without robotic assistance for 1 hour every day for 3 weeks.
  Other Names: WALK
  Arms: Walking training
Other: Control group — The control group performed the physiotherapy treatment for 3 weeks.
  Other Names: CON
  Arms: Control group

SUMMARY:
We are conducting a three-group comparative study on stroke patients. The treatment is started in a subacute state and completed in the hospital. The essence of robot-assisted treatments is faster recovery and better learning to walk. The group will do a special walking exercise with a robot. The walking group does the same training, only without robotic assistance. The control group will receive physiotherapy treatments financed by the state. Control examination after 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

post stroke 6MWT : 120> minimum after stroke 3 days be a stroke patient first stroke hemiplegia

Exclusion Criteria:

multiple strokes, inability to stand and walk, cognitive function disorder does not reach 50 meters with a minimal walking aid Alcohol Sever heart problem sever demeanor alcoholism drug problems Drug

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-09 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 3 weeks (0-5 score, high score better)
  stroke, diagnostic, quality of life

SECONDARY OUTCOMES:
Barthel Index for Activities of Daily Living (ADL) | 3 weeks
  stroke quality of life
Berg Balance Scale | 3 weeks (0-30, high score better)
  balance test
10-m maximal walking speed | 3 weeks
  high speed test
6MWT | 3 weeks
  walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Tollár József, Kaposvár, Somogy County, Hungary

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=soft%20exoskeleton&page=3